CLINICAL TRIAL: NCT05184959
Title: Correlation Between Early Neuro-immune Metabolism in Patients With Benzodiazepine Poisoning and Mental Disorders With Depression --- A Multiple Center Observational Study
Brief Title: Correlation Between Immune Metabolism in Patients With Benzodiazepine Poisoning and Patients'Mental Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1069
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Poisoning by Benzodiazepines; Depression
Keywords: poisoning; benzodiazepines; neuro-immunity
MeSH Terms: conditions — Depression; Poisoning

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — serum obtained by centrfuge
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
High-dose benzodiazepines can inhibit the central nervous system, respiratory system and cardiovascular motor center, resulting in loss of consciousness, disappearance of reflex, respiratory inhibition, decrease of blood pressure and so on. This kind of drug acute poisoning is the most common drug poisoning in internal medicine. It has acute onset and severe symptoms. If it is not treated properly in time, it can be life-threatening. At present, the research on the accumulation and metabolic state caused by benzodiazepine poisoning is not sufficient; at the same time, the changes of neuroendocrine metabolism and immune function of patients with neuroendocrine metabolism and immune function need to be further explored. Therefore, the main purpose of this study is to analyze the effects of neuroendocrine metabolism and immune function on organ function and mental state in patients with benzodiazepine poisoning.

DETAILED DESCRIPTION:
Benzodiazepines are the first choice for clinical anti-anxiety, sedation and hypnosis, as well as anticonvulsant, antiepileptic and central muscle relaxation. Commonly used are diazepam (diazepam), nitro diazepam, clonazepam, alprazolam, triazolam and so on. The drug itself is an inhibitor of the central nervous system, which has a high selectivity for the inhibition of the central nervous system, mainly inhibiting the limbic system of the brain and less inhibitory effect on the reticular ascending activation system. It mainly acts on the synaptic sites of GABA-Ergic nerve endings in the central nervous system. It enhances the affinity between GABA and its receptors by binding to benzodiazepine receptors, thus increasing the open frequency of Cl- channels coupled with GABA receptors and exerting an inhibitory effect. High-dose benzodiazepines can inhibit the central nervous system, respiratory system and cardiovascular motor center, resulting in loss of consciousness, disappearance of reflex, respiratory inhibition, decrease of blood pressure and so on. This kind of drug acute poisoning is the most common drug poisoning in internal medicine. It has acute onset and severe symptoms. If it is not treated properly in time, it can be life-threatening. At present, the research on the accumulation and metabolic state caused by benzodiazepine poisoning is not sufficient; at the same time, the changes of neuroendocrine metabolism and immune function of patients with neuroendocrine metabolism and immune function need to be further explored. Therefore, the main purpose of this study is to analyze the effects of neuroendocrine metabolism and immune function on organ function and mental state in patients with benzodiazepine poisoning.

ELIGIBILITY:
Inclusion Criteria:

Benzodiazepine poisoning Within 6 hours, at least one target organ dysfunction. No bad habits (drug use, alcohol addiction)

Exclusion Criteria:

Refusal to join this study Lack of information/incompleteness Vulnerable groups such as pregnant women, incapable of civil conduct and indeterminate agent consent Chronic multiple organ dysfunction Tumors, blood system diseases, various systemic immune diseases Various infectious diseases (various hepatitis, tuberculosis, AIDS)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: posioning with Benzodiazepine along with at least one organ dysfucntion
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Time interval | at admittion
  Interval from benzodiazepine poisoning to emergency pre-examination